CLINICAL TRIAL: NCT00733629
Title: In Vitro Studies pf Endothelial Cells Derived From HHT Patients
Brief Title: Study of Endothelial Cells in Patients With Hereditary Haemorrhagic Telangiectasia
Status: Withdrawn | Type: Observational
Why Stopped: Technical reasons- unable to process samples therefore did not recruit
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IC/CLS4
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endothelial cells

SUMMARY:
Hereditary Haemorrhagic Telangiectasia (HHT, also known as Osler-Weber-Rendu Syndrome) is an disease that leads to the development of dilated and fragile blood vessels. We propose to culture endothelial cells from patients with HHT, to culture cells that express the proteins mutated in HHT, namely endoglin and ALK-1. We will study the properties of these cells which will involve their growth in different conditions and anticipate that DNA, mRNA and proteins will be extracted from these cells for study of cell responses and association with expression levels of endoglin and ALK-1. We hypothesize that these cells which express "half-normal" endoglin or ALK-1 will show altered protein synthetic differences when compared to normal white blood cells. We anticipate that that these findings may help to explain aspects of the HHT disease phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hereditary haemorrhagic telangiectasia and family members

Exclusion Criteria:

* Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hereditary haemorrhagic telangiectasia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2002-08; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith Campus, London, United Kingdom